CLINICAL TRIAL: NCT04959097
Title: Retinoblastoma Patient Clinical Database, Liquid Biopsy and Tissue Biorepository
Brief Title: RB Liquid Biopsy Biorepository
Acronym: rbliqbx
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Jesse Berry, Associate Professor of Ophthalmology, Children's Hospital Los Angeles
Other Study IDs: CHLA-17-00248
Record Dates: First submitted 2021-06-24; First posted 2021-07-13 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Retinoblastoma; Retinoblastoma Bilateral; Retinoblastoma Unilateral
Keywords: Retinoblastoma; RB; Ocular oncology; Aqueous humor
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Aqueous Humor, Blood, Saliva, Tumor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retinoblastoma (RB) is a primary eye cancer that forms in the back of the eye of infants and toddlers. Traditionally, RB is diagnosed without a biopsy; tumor can only be studied once an eye has been surgically removed.

Given this limitation, we use aqueous humor (AH), the clear fluid in the front of the eye to detect specific markers, or information, that comes from the tumor itself.

DETAILED DESCRIPTION:
Retinoblastoma (RB) is a primary intraocular malignancy that forms in the retina of infants and toddlers. Traditionally, RB is diagnosed without tissue as direct tumor biopsy is prohibited due to risk of extraocular spread; tissue can only be obtained once an eye has been surgically removed.

Given this limitation, there are no eye-specific molecular biomarkers in current clinical practice for RB. The lack of in vivo molecular data without removing the eye limits our ability to prognosticate clinical outcomes and develop personalized treatment plans. It also limits our understanding of intratumoral dynamics throughout therapy.

The aqueous humor (AH) is a high-yield source of tumor-derived nucleic acid that can be utilized as a liquid biopsy in eyes with retinoblastoma. Detection of biomarkers from the AH may be used to prognosticate the likelihood of eye salvage and in the future may facilitate targeted, patient-centered therapies based on molecular biomarkers.

OBJECTIVES:

1. Systematically and prospectively record accurate and complete data regarding the clinical presentation, treatment, and outcomes of patients diagnosed with RB.
2. Collect, bank, preserve, and analyze biomaterials including AH, blood and saliva from patients with RB.
3. Correlate phenotypic data with genotypic findings from human biomaterials in retinoblastoma patients to identify clinically relevant biomarkers

ELIGIBILITY:
Inclusion Criteria:

* All patients, age 0 days to 18 years, with a diagnosis unilateral or bilateral retinoblastoma (RB) seen at CHLA (Children's Hospital Los Angeles).

Exclusion Criteria:

* Patients referred for second opinions only and not treated at CHLA for any reason.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients, age 0 days to 18 years, with a diagnosis unilateral or bilateral retinoblastoma (RB) treated at CHLA who have biospecimens taken for research during the course of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of Ocular Salvage (eye saved) with biomarkers | through study completion, a minimum of 12 months after diagnosis and average of 24 months
  We aim to evaluate whether any identifiable molecular biomarkers (e.g. chromosomal alterations or tumor fraction) in the aqueous or blood can predict ocular salvage, or the likelihood of saving the eye with therapy
Identification of RB1 (RB Transcriptional Corepressor 1) gene mutations from the AH liquid biopsy | through study completion, a minimum of 12 months after diagnosis and average of 24 months
  We aim to identify both somatic and germline RB1 gene mutations in the AH

SECONDARY OUTCOMES:
Correlation of High-Risk Histopathologic Features with presence of biomarkers | through study completion, a minimum of 12 months after diagnosis and average of 24 months (only if the eye is enucleated)
  We aim to evaluate whether any identifiable molecular biomarkers in the aqueous or blood can predict the presence of high risk histopathologic features that are known to increase risk of metastatic disease
Correlation of class of Seeding with presence of biomarkers | through study completion, a minimum of 12 months after diagnosis and average of 24 months
  We aim to evaluate whether any identifiable molecular biomarkers in the aqueous or blood are associated with the presence of type of seeding

CONTACTS AND LOCATIONS:
Overall Officials: Jesse L Berry, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available to other researchers via NIH GDS/dbGAP controlled databases.
Time Frame: October 2023
URL: https://www.ncbi.nlm.nih.gov/gap/

REFERENCES:
- [Background] Berry JL, Xu L, Murphree AL, Krishnan S, Stachelek K, Zolfaghari E, McGovern K, Lee TC, Carlsson A, Kuhn P, Kim JW, Cobrinik D, Hicks J. Potential of Aqueous Humor as a Surrogate Tumor Biopsy for Retinoblastoma. JAMA Ophthalmol. 2017 Nov 1;135(11):1221-1230. doi: 10.1001/jamaophthalmol.2017.4097. PMID 29049475
- [Background] Berry JL, Xu L, Polski A, Jubran R, Kuhn P, Kim JW, Hicks J. Aqueous Humor Is Superior to Blood as a Liquid Biopsy for Retinoblastoma. Ophthalmology. 2020 Apr;127(4):552-554. doi: 10.1016/j.ophtha.2019.10.026. Epub 2019 Oct 31. PMID 31767439
- [Result] Berry JL, Xu L, Kooi I, Murphree AL, Prabakar RK, Reid M, Stachelek K, Le BHA, Welter L, Reiser BJ, Chevez-Barrios P, Jubran R, Lee TC, Kim JW, Kuhn P, Cobrinik D, Hicks J. Genomic cfDNA Analysis of Aqueous Humor in Retinoblastoma Predicts Eye Salvage: The Surrogate Tumor Biopsy for Retinoblastoma. Mol Cancer Res. 2018 Nov;16(11):1701-1712. doi: 10.1158/1541-7786.MCR-18-0369. Epub 2018 Jul 30. PMID 30061186
- [Result] Xu L, Polski A, Prabakar RK, Reid MW, Chevez-Barrios P, Jubran R, Kim JW, Kuhn P, Cobrinik D, Hicks J, Berry JL. Chromosome 6p Amplification in Aqueous Humor Cell-Free DNA Is a Prognostic Biomarker for Retinoblastoma Ocular Survival. Mol Cancer Res. 2020 Aug;18(8):1166-1175. doi: 10.1158/1541-7786.MCR-19-1262. Epub 2020 May 20. PMID 32434859
- [Result] Xu L, Shen L, Polski A, Prabakar RK, Shah R, Jubran R, Kim JW, Biegel J, Kuhn P, Cobrinik D, Hicks J, Gai X, Berry JL. Simultaneous identification of clinically relevant RB1 mutations and copy number alterations in aqueous humor of retinoblastoma eyes. Ophthalmic Genet. 2020 Dec;41(6):526-532. doi: 10.1080/13816810.2020.1799417. Epub 2020 Aug 17. PMID 32799607
- [Result] Polski A, Xu L, Prabakar RK, Kim JW, Shah R, Jubran R, Kuhn P, Cobrinik D, Hicks J, Berry JL. Cell-Free DNA Tumor Fraction in the Aqueous Humor Is Associated With Therapeutic Response in Retinoblastoma Patients. Transl Vis Sci Technol. 2020 Sep 30;9(10):30. doi: 10.1167/tvst.9.10.30. eCollection 2020 Sep. PMID 33062393
- [Result] Xu L, Kim ME, Polski A, Prabakar RK, Shen L, Peng CC, Reid MW, Chevez-Barrios P, Kim JW, Shah R, Jubran R, Kuhn P, Cobrinik D, Biegel JA, Gai X, Hicks J, Berry JL. Establishing the Clinical Utility of ctDNA Analysis for Diagnosis, Prognosis, and Treatment Monitoring of Retinoblastoma: The Aqueous Humor Liquid Biopsy. Cancers (Basel). 2021 Mar 13;13(6):1282. doi: 10.3390/cancers13061282. PMID 33805776